CLINICAL TRIAL: NCT05591287
Title: Contrast Enhanced Harmonic Endoscopic Ultrasound (CH-EUS), Elastography, and Fractal Analysis in Predicting Pancreatic Cancer Aggressiveness and Response to Therapy.
Acronym: CH-E-EUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3251
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Mass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Contrast enhanced harmonic Endoscopic Ultrasound — Solid pancreatic masses suspected for PDAC detected by cross-sectional imaging and confirmed at EUS will be enrolled. The

SUMMARY:
Contrast enhanced harmonic Endoscopic Ultrasound (CH-EUS) can be used during a conventional EUS examination to correctly identify and target lesions with the help of Ultrasound Contrast Agents. When CH-EUS is applied to the dynamic ultrasound images of conventional EUS, additional information about tumour vascularity can be obtained solely from the visual uptake of contrast agent into the tumour. Angiogenesis within malignant tumour tissue is varied from that of its normal surrounding tissue.Blood flow within malignant tissue is characteristically low volume. Contrast agents are slow to pass through tumour microvasculature and hence this is seen as an area of hypo-enhancement. This hypo-enhancement or hypo-vascularity is well demonstrated in PDAC and the opposite is known to be true for PNET, both of these findings showing to be consistent with cytopathological results.Tumour hemodynamics and vascular patterns resultant from contrast uptake can be analysed further with the help of fractal use. Attaining this information can allow more accurate characterization of both PDAC and PNET thus in turn predicting their respective behaviours i.e., aggressiveness (local or systemic spread) and histological grade. (6)

Contrast-enhanced computer tomography (CT) is currently used to evaluate the response of chemotherapy in patients with PDAC according to the RECIST guidelines. However, one significant advantage of CH-EUS over dynamic CT imaging is that ultrasound contrast agents do not leak into the interstitial space allowing for better quantitative measurement of tissue perfusion.More recently, the EFSUMB guidelines have recommended dynamic CH-EUS as a preferred technique to monitor anti-angiogenic treatment.This founds the basis for evaluating CH-EUS's role. *(with the help of fractal analysis)-remove this if needed* in predicting PDAC's response to neo-adjuvant chemotherapy as this is yet to be evaluated.

Yamashita et al. demonstrated that patients with PDAC with positive vessel sign showed a significantly longer progression free survival compared with patients with negative vessel sign after chemotherapy (P = 0.037; log-rank test).

EUS elastography (EUS-E) is a US technique that measures the hardness of tissues. The level of hardness of SPLs can be evaluated using qualitative scores and/or quantitative methods (strain ratio [SR]).

ELIGIBILITY:
Inclusion Criteria:

* Patients>18 years old.
* Solid pancreatic masses suspected for PDAC detected by cross-sectional imaging and confirmed at EUS will be enrolled. The exclusion criteria will be: patients who decline to participate in the study, patients with contraindication to the procedure.

Exclusion Criteria:

* Contra-indication to Sonovue (allergic reaction, uncontrolled hypertension, pulmonary hypertension, previous episode of acute coronary syndrome or documented coronary artery disease, heart failure, arythmia)
* pregnancy
* lactating mothers
* severity of disease
* presence of cyst volume of > 25% of the total volume of the lesion
* patients who decline to participate in the study
* patients with contraindication to the procedure.
* Patients who had received previous chemotherapy or radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid pancreatic masses suspected for PDAC detected by cross-sectional imaging and confirmed at EUS will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor aggressiveness | 2 years
  To identify the correlation between the CH-EUS, elastography, and fractal-based analysis, and pancreatic cancer aggressiveness. grading is expressed from the pathological analysis of the resected specimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No